CLINICAL TRIAL: NCT04180111
Title: Cross Linking Corneal Biomechanical Evaluation of CATS Tonometer Prism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Intuor Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CATS crosslink
Record Dates: First submitted 2019-11-23; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: CATS Tonometer — CATS Tonometer Prism

SUMMARY:
The purpose of this study is to determine if the device, CATS tonometer prism, measures intraocular pressure significantly differently than the current standard of care tonometer prism (Goldmann) before and after a corneal crosslinking procedure. This difference would be a measurement of the amount of corneal biomechanical changes made due to the cross-linking procedure.

DETAILED DESCRIPTION:
This clinical trial is a prospective, controlled, study and will be performed at one clinical investigative sites in Tucson Arizona1. The purpose of this study is to determine if the device, CATS tonometer prism, measures intraocular pressure significantly differently than the current standard of care tonometer prism (Goldmann) before and after a corneal crosslinking procedure. This difference would be a measurement of the amount of corneal biomechanical changes made due to the cross-linking procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, at least 18 years of age
* Subject has a clear understanding and agrees to all the conditions of the informed consent form

Exclusion Criteria:

* • Subject has undergone ocular surgery within the last 3 months

  * Uncontrolled systemic disease that in the opinion of the Investigator would put the subject's heath at risk
  * Pregnant or nursing women
  * Those who have had corneal surgery including corneal laser surgery
  * Microphthalmos
  * Buphthalmos
  * Severe Dry eyes
  * Lid squeezers - blepharospasm
  * Nystagmus
  * corneal or conjunctival infection.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty three (23) Subjects 18 years and older and will be enrolled from one clinical. Subjects will be chosen from patients who are being examined for a corneal cross-linking procedure.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2019-05-05 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
IOP measurement | 6 months
  comparative IOP measurement between CATS and GAT tonometer prisms

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona Eye Consultants, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided